CLINICAL TRIAL: NCT02597348
Title: Curative Potential of Liver Transplantation in Patients With Definitively Unresectable Colorectal Liver Metastases (CLM) Treated by Chemotherapy: a Prospective Multicentric Randomized Trial
Brief Title: Liver Transplantation in Patients With Unresectable Colorectal Liver Metastases Treated by Chemotherapy
Acronym: TRANSMET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P130922
Record Dates: First submitted 2015-10-23; First posted 2015-11-05 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Liver Metastasis; Colorectal Cancer; Metastasis
Keywords: Liver; Metastasis; Colorectal cancer; Liver transplantation
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liver Transplantation (Experimental): Arm LT+C: patients will be treated by experimental liver transplantation preceding the non experimental standard chemotherapy (according to usual practices).
  Interventions: Procedure: Liver Transplantation
- No intervention (No Intervention): Arm C: patients will receive non experimental standard chemotherapy according to usual practices in the context of definitively unresectable CLM.

INTERVENTIONS:
Procedure: Liver Transplantation — The patient of the arm LT+C are treated by experimental liver transplantation preceding the Non experimental standard chemotherapy (according to usual practices) .
  Other Names: Experimental LT+Non Experimental Usual Chimiotherapy
  Arms: Liver Transplantation

SUMMARY:
This is a multicentric randomized parallel group open trial comparing 5-year survival of chemotherapy followed by LT (Group LT+C) versus chemotherapy alone (Group C) in patients with confirmed unresectable liver-only metastases, well controlled by chemotherapy (no progression) and extensively explored by modern imaging techniques. The primary objective of the trial is to validate in a large multicentric cohort of selected patients the possibility to obtain at least 50% 5-years survival with LT combined to chemotherapy compared to around 10% with chemotherapy alone.

DETAILED DESCRIPTION:
Liver transplantation (LT) has recently been proposed as alternative treatment for definitively unresectable colorectal liver metastases in selected patients with a 60% estimated survival at 5 years in a recent prospective Norwegian study. However, disease free survival (DFS) in this preliminary study has been poor with 90% of recurrence after LT.

The objective of our study is to validate LT as a therapeutic option on a large multicentric scale throughout a highly strict policy selection in term of survival, disease free survival and quality of life. In order to reduce selection bias, unresectability criteria and theorical indication to LT will be confirmed by an independent Steering Committee including HPB surgeons, oncologists, radiologists and hepatologists.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 65 years
* Good performance status, ECOG 0 or 1 (39).
* Histologically proved adenocarcinoma in colon or rectum
* BRAF wild-type CRC on primary tumor or liver metastases
* High standard oncological surgical resection of the primary defined by :

  * Safe margin of resection
  * Curative resection of primary tumor according to oncological principles
  * TNM adequate staging
* Absence of local recurrence on colonoscopy performed in the 12 months prior to inclusion (except in case of primary tumor resection < 12 months )
* Confirmed non resectable colorectal liver metastases by the validation committee
* ≥ 3 months of tumor control during the last chemotherapy line: Stable or Partial Response on RECIST criteria (40)
* ≤ 3 lines of chemotherapy for metastatic disease
* CEA < 80 microg/L or a decrease ≥ 50% of the highest serum CEA levels observed during the disease
* Absence of extrahepatic tumor localisation according to CT scan and PET-CT
* Renal function should be within the normal limits
* No need for extra-renal purification procedure, hemodialysis or kidney transplantation associated (nephrologist assessment)
* A platelet count> 80,000 / mm3
* White blood cell count> 2500 / mm3
* Eligible for both treatments groups
* Signed informed consent and expected cooperation of the patient for the treatment and follow up

Exclusion Criteria:

* Participation refusal
* No health insurance facilities
* General contraindication to LT (Severe cardiopulmonary disease or other life-limiting coexisting medical conditions, extrahepatic malignancy, active alcohol or substance abuse, active infection or uncontrolled sepsis, lack of psychosocial support or inability to comply with medical treatment)
* Other malignancies either concomitant or within 5 years before liver transplantation
* Patients not having received standard treatment for the primary CRC according to recommended guidelines
* Prior extra hepatic metastatic disease or local relapse
* Pregnancy at the time of inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
5 years overall survival (OS) | 5 years
  The evaluation of 5-years overall survival will be conducted by constructing survival curves using the Kaplan-Meier method. Graphs will be created following the best practices defined by Pocock.
  * If the proportionality of hazards is respected: Survival in each randomization arm will be compared using the Log-Rank test. The hazard ratio and the associated 95% confidence interval will be estimated using a Cox proportional hazards model.
  * If the proportionality of hazards is not respected: the difference in Restricted Mean Survival Time (RMST) between the arms and the associated 95% confidence interval will be estimated.
  The randomization stratification by cluster of centers will not be taken into account in the analyses. This is because it was done for administrative reasons.

SECONDARY OUTCOMES:
3-years overall survival (OS) | 3 years
Disease free survival (DFS) (Arm LT+C) or Progression free survival (PFS) (Arm C) | 3 and 5 years
Recurrence rate at 3 and 5 years | 3 and 5 years
  Radiological assessment will be performed according to the RECIST criteria and confirmed by 2 local radiologists.
Quality of life (QOL) of patients using the European Organization for Research and Treatment of Cancer (EORTC) questionnaires.: QLQ-C30 | year 5
  QLQ-C30 covers general aspects of health-related quality of life
Quality of life (QOL) of patients using the European Organization for Research and Treatment of Cancer (EORTC) questionnaires.: QLQ-LMC21 | year 5
  QLQ-LMC21 is valid and reliable questionnaire module to use with the QLQ-C30 in assessing in hepatectomy or palliative treatment for colorectal liver metastases
Quality of life (QOL) of patients of Group LT followed by chemotherapy, using the NIDDK questionnaire of Liver Transplantation Database | year 5

CONTACTS AND LOCATIONS:
Overall Officials: René ADAM, PhD, Principal Investigator — AP-HP, Paul Brousse Hospital
Locations (1):
- AP-HP, Paul Brousse Hospital, Villejuif, France

REFERENCES:
- [Derived] Adam R, Piedvache C, Chiche L, Adam JP, Salame E, Bucur P, Cherqui D, Scatton O, Granger V, Ducreux M, Cillo U, Cauchy F, Mabrut JY, Verslype C, Coubeau L, Hardwigsen J, Boleslawski E, Muscari F, Jeddou H, Pezet D, Heyd B, Lucidi V, Geboes K, Lerut J, Majno P, Grimaldi L, Levi F, Lewin M, Gelli M; Collaborative TransMet group. Liver transplantation plus chemotherapy versus chemotherapy alone in patients with permanently unresectable colorectal liver metastases (TransMet): results from a multicentre, open-label, prospective, randomised controlled trial. Lancet. 2024 Sep 21;404(10458):1107-1118. doi: 10.1016/S0140-6736(24)01595-2. PMID 39306468

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT02597348/SAP_000.pdf